CLINICAL TRIAL: NCT02034175
Title: Comparison of the Somnarus Sleep Apnea Diagnostic Technology SomnaPatch With Polysomnography in Sleep Disordered Breathing
Brief Title: Comparison of SomnaPatch With Polysomnography in Sleep Disordered Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somnarus Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: SomnaPatch-001-D
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea; Central Sleep Apnea; Mixed Sleep Apnea; Cheyne-Stokes Respiration
Keywords: apnea; hypopnea; polysomnography; respiratory; cheyne
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea, Central; Sleep Apnea Syndromes; Cheyne-Stokes Respiration; Apnea | interventions — Polysomnography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The two sets of data (PSG and Somnapatch) were scored independently. Therefore it was masked what set of data belonged to what individual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SomnaPatch (Experimental): SomnaPatch is a standalone flexible diagnostic skin-adhesive patch with electronics inside. The patch is placed on the patient's face.
  Interventions: Device: SomnaPatch
- Polysomnography (Active Comparator): Polysomnography performed in a sleep lab is considered a gold standard in diagnosing the sleep breathing disorders.
  Interventions: Device: Polysomnography

INTERVENTIONS:
Device: SomnaPatch — SomnaPatch is a standalone flexible diagnostic skin-adhesive patch with electronics inside. The patch is placed on the patient's face.
  Arms: SomnaPatch
Device: Polysomnography — Polysomnography performed in a sleep lab is considered a gold standard in diagnosing the sleep breathing disorders.
  Arms: Polysomnography

SUMMARY:
The purpose of this study is to evaluate the accuracy of Somnarus diagnostic technology for diagnosis of sleep apnea in human subjects. This includes evaluation of Somnarus technology in Obstructive Sleep Apnea (OSA) and Central Sleep Apnea (CSA), including Cheyne - Stokes respiration (CSR).

DETAILED DESCRIPTION:
This is a multi- center, open label study to evaluate the accuracy of Somnarus device when compared with overnight polysomnographic measurements.

The study includes the following steps:

Screening the database or advertising among cardiologists, neurologists, pulmonologists and Ear Nose and Throat (ENT) specialists to identify potential subjects.

Initial visit, includes:

1. Consent discussion and signature
2. History, vital signs, and physical exam

Night study

a. A polysomnogram is conducted and, at the same time, a SomnaPatch device is used.

Additional visits If side effects occur, or if the data collection fails, or at the request of the sponsor to repeat the sleep study for further data collection and comparison.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign the informed consent
* Able to comply with visits and follow ups included in this protocol
* Ages 20-85 years

Exclusion Criteria:

* An unstable medical condition, acute or chronic, that in the opinion of the investigator puts the subject at health risks related this trial or interferes with the clinical trial and data collection.
* Skin rash on the nose or on the maxillary area.
* A history of skin allergy to medical tape, and hypoallergenic tapes.
* A history of skin cancer on the nose or on the maxillary area.
* A history of the base of skull fractures, facial fractures

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merhan Farid-Moayer, MD, Principal Investigator — Peninsula Sleep Center
Locations (3):
- United States (3):
  - Preferred Research Partners, Inc, Little Rock, Arkansas
  - Peninsula Sleep Center, Burlingame, California
  - The Good Sheperd Sleep Center, LLC, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multi-site study conducted in the United States. Study enrollment began February 2016 and concluded November 2016.
Groups:
- SomnaPatch and PSG Simultaneously: All patients enrolled in the clinical trial underwent simultaneous testing with both polysomnography and SomnaPatch portable sleep monitor
Period: Overall Study
Arm/Group | SomnaPatch and PSG Simultaneously
Started | 190
Completed | 190
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SomnaPatch and PSG Simultaneously
Number analyzed (Participants) | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 172
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 146
  More than one race | 7
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 190

OUTCOME MEASURES:

1. Primary Outcome: Agreement Between Polysomnography (PSG) and SomnaPatch in Detecting Patients Apnea-Hypopnea Index (AHI)
Description: AHI is the number of apneas and hypopneas that occur over an hour during the course of the night. The SomnaPatch and PSG were wore simultaneously over the night. The results from the SomnaPatch and PSG were compared per individual for agreement
Time Frame: 1 night
Population: 12 participants were excluded due to poor quality of sleep data or technical issues during the night. Sleep data was unable to be scored.
Measure: Number (95% Confidence Interval); unit: percentage of device agreements
Arm/Group | SomnaPatch and PSG Simultaneously
Number analyzed (Participants) | 178
percentage of device agreements | 87.1 [81.2 to 91.6]

ADVERSE EVENTS:
Time Frame: All adverse events were collected over the 1 night period
Arm/Group | SomnaPatch and PSG Simultaneously
All-Cause Mortality (participants affected / at risk) | 0/190
Serious Adverse Events (participants affected / at risk) | 0/190
Other Adverse Events (participants affected / at risk) | 0/190

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is responsible for publishing the study results and the PIs are not allowed to publish the study data without an approval from the sponsor